CLINICAL TRIAL: NCT02757456
Title: Aerobic Exercise and Vascular Hemodynamic Parameters Among Prevalent Hemodialysis Population
Brief Title: Exercise and Vascular Parameters in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sameena Iqbal (Other)
Responsible Party: Sponsor-Investigator, Sameena Iqbal, MD FRCP MSc., McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-309-GEN
Record Dates: First submitted 2012-11-19; First posted 2016-05-02 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2016-04

CONDITIONS: Cardiovascular Disease
Keywords: exercise; hemodialysis; pulse wave velocity; micro RNAs
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Exercise program (Other): Intervention of aerobic exercise
  Interventions: Behavioral: Aerobic Exercise program
- Control (Other): no aerobic exercise program
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Aerobic Exercise program — The 16-week program will consist of aerobic-type steady-state or interval exercises using a pedals attachable to the dialysis chairs. The purpose will be to slowly increase exercise duration by 5 minute increments to reach the goal of 30 min/treatment. The exercise program during hemodialysis sessions will contain a combination of aerobic and flexibility exercises, about 30 minutes of cycling with 10 minutes of warm up/stretching exercises and 10-15 minutes cool down. The frequency of exercise will be three sessions a week, during the first hour of dialysis treatment for the duration of 16 weeks. Blood pressure and heart continuous monitoring will be carried out during the exercise program. Exercise log sheets will be filled for each session for the 16 weeks.
  Arms: Aerobic Exercise program
Other: Control — No aerobic exercise is offered but baseline and end of study testing of the outcomes occur
  Arms: Control

SUMMARY:
Arterial calcification is very common in the incident hemodialysis population, ranging 71-83%.Given that cardiovascular disease is a major cause of mortality in the hemodialysis population, medial arterial calcification may contribute through increased risk of sudden death and congestive heart failure. Applanation tonometry is the method of choice to measure pulse wave velocity and pulse wave analysis. The primary objective will be to assess the effect of a 16 week exercise program on aortic pulse wave velocity as the vascular parameter and gait speed as the physical functioning parameter. The secondary objectives will assess the effect of the exercise program on ultrafiltration rates, weight, SBP, DBP, BNP, hsTroponin, serum calcium, phosphate, albumin, glucose, LDL, HDL, TG, glycated hemoglobin, hemoglobin, CRP, micro RNAs (21, 126, 133, 146a, 221/222 and 210) and hospitalizations.

DETAILED DESCRIPTION:
The investigators propose a pilot project to assess the effect of a 16 week aerobic exercise program on arterial stiffness and cardiovascular risk in the hemodialysis population. The primary objective will be to assess the effect of a 16 week exercise program on aortic pulse wave velocity as the vascular parameter and gait speed as the physical functioning parameter. The secondary objectives will assess the effect of the exercise program on ultrafiltration rates, weight, SBP, DBP, BNP, hsTroponin, serum calcium, phosphate, albumin, glucose, LDL, HDL, TG, glycated hemoglobin, hemoglobin, CRP, micro RNAs (21, 126, 133, 146a, 221/222 and 210) and hospitalizations.

Study Design:

Randomized-controlled study of end stage renal disease patients between the age of 18 and 90 years to assess the effect of exercise on arterial stiffness. Our aim is to have 23 patients in both groups. The study period will be 24 weeks-4 weeks for recruitment, 16 weeks for the intervention and 4 weeks for data collection and analysis. The protocol will be submitted to the MUHC Research Ethics Board.

The following outcomes are of interest:

1. change in gait speed before and after the exercise program
2. change in pulse wave velocity before and after the exercise program
3. change in BNP, blood pressure, dialysis ultrafiltration, hemoglobin, micro RNAs before and after the exercise program

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-95 years
2. Able to comply with the study procedures and medication
3. Written informed consent given
4. On a stable in-center hemodialysis regimen (at least 3 times per week) for ≥ 12 weeks prior to recruitment
5. Cardiac evaluation within the year with adequate cardiac function to be able to undergo the exercise program

Exclusion Criteria:

1. Participation in any clinical trial using an investigational product or device during the 30 days preceding recruitment
2. Any physical or psychological disability that would impact study participation, such as severe cerebrovascular disease (ie. hemiparesis, cerebellar ataxia, etc.) or dementia
3. Serum iPTH > 250 pmol/L within 30 days prior to screening visit
4. Dysrhythmia or severe cardiac disease: CHF Class III-IV; unstable cardiovascular diagnosis (for example MI, CABG, PTCA, CVA, and TIA) within 90 days prior to recruitment
5. Severe peripheral vascular disease
6. Severe hyperkalemia (>6.5 mmol/L) consistently for the last 2 weeks
7. Current active cancer (excluding basal cell carcinoma of the skin)
8. Poorly controlled hypertension (systolic > 180mmHg or diastolic > 100mmHg) within 4 weeks prior to recruitment
9. Anticipated live donor kidney transplant or any other planned major surgery over the study duration
10. History of poor adherence to hemodialysis or medical regimen
11. Any disease or condition, physical or psychological that, in the opinion of the investigator, would compromise the safety of the subject or the likelihood of achieving reliable results or increase the likelihood of the subject being withdrawn

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Gait speed | at 24 weeks and 48 weeks
  The gait speed will be measured with a timer (in seconds) as the subject will be asked to walk a 10 foot or 3 meter course and back as quickly as possible. Two readings will be taken and the average will be recorded.

SECONDARY OUTCOMES:
Change from Baseline Pulse wave velocity (PWV) | at 24 weeks and 48 weeks
  PWV measurements will be performed between the carotid and femoral artery sites, to primarily measure the stiffness of the aorta. A 3-lead ECG will be used in conjunction with a tonometer to measure the pressure pulse waveform sequentially in the two peripheral artery sites
Change from Baseline Pulse wave analysis | at 24 and 48 weeks
  Wave Reflections and Arterial Stiffness. Analysis of the systolic part of the central pressure waveform will be performed to evaluate PWV and the LV afterload. The main indices that were described above (in hemodynamic measurements) will be obtained by aortic PWA.
Change from baseline Rand survey | at 24 weeks and 48 weeks
  RAND 36-item survey will be used to assess physical functioning and fatigue. This survey has been validated in the Hemodialysis population. The survey consists of 36 items and takes approximately 5-10 minutes to complete.

OTHER OUTCOMES:
change from baseline micro RNA levels | at 24 weeks and 48 weeks
  micro RNAs (21, 126, 133, 146a, 221/222 and 210): blood sample will be taken before initiation of dialysis week of baseline measurements and end of study.
change from baseline Brain Natuiretic Peptide | at 24 weeks and 48 weeks
  Brain Natuiretic Peptide: measure before initiation of dialysis at baseline and at the end of study period.
change from baseline troponin levels | at 24 weeks and 48 weeks
  to assess myocardial injury during dialysis at baseline and at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Sameena Iqbal, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No